CLINICAL TRIAL: NCT02301676
Title: Phase 4 Study of Long Term Postoperative Cognitive Dysfunction After Laparoscopic Cholecystectomy in the Elderly Patients
Brief Title: Long Term Postoperative Cognitive Dysfunction in the Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Eun-Jung Kim, anesthesiologist, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LPOCD60
Record Dates: First submitted 2014-10-08; First posted 2014-11-26 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Cognitive Impairment
Keywords: Geriatrics; Cognitive impairment; Interviews, Telephone
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia & Control (Active Comparator): After the surgery, the patients are discharged from the hospital, investigators will check the postoperative cognitive function 4 times: 1weak, 3months, 6months, 1 year later using the intervention "Korean version of telephone interview for cognitive status (TICS)". The test will be administered to spouse simultaneously by telephone.
  Interventions: Behavioral: Korean version of telephone interview for cognitive status
- Sevoflurane & Propofol & Dexmedetomidine (Active Comparator): The anesthetic methods are divided into the following 3 kinds: Sevoflurane, Propofol, Dexmedetomidine. These anesthetic drugs are used in general anesthesia generally.
  Interventions: Drug: Sevoflurane; Drug: propofol; Device: dexmedetomidine

INTERVENTIONS:
Behavioral: Korean version of telephone interview for cognitive status — The telephone interview for cognitive status (TICS), developed by Brandt et al. (1988), is one of the most popular telephone interview-based screening instruments. Especially, the Korean version of TICS is translated more suitable for Korean culture with the permission of the authors of the original version. The Korean version of TICS consists of 11 items, total score is 41.
  Other Names: TICS
  Arms: General anesthesia & Control
Drug: Sevoflurane — Sevoflurane is one of the most commonly used volatile anesthetic agents, particularly for outpatient anesthesia, and including in anesthesia of children and infants, and in veterinary medicine.
  Other Names: sevofrane
  Arms: Sevoflurane & Propofol & Dexmedetomidine
Drug: propofol — Propofol is highly protein-bound in vivo and is metabolized by conjugation in the liver. The half-life of elimination of propofol has been estimated to be between 2 and 24 hours.
  Other Names: fresofol
  Arms: Sevoflurane & Propofol & Dexmedetomidine
Device: dexmedetomidine — Dexmedetomidine is a sedative medication used by intensive care units and anesthesiologists. It is relatively unusual in its ability to provide sedation without causing respiratory depression.
  Other Names: precedex
  Arms: Sevoflurane & Propofol & Dexmedetomidine

SUMMARY:
The purposes of this study are to determine whether long-term postoperative cognitive dysfunction (POCD) is occured after general anesthesia and anesthetic drugs have an effect on the result about POCD.

DETAILED DESCRIPTION:
In present aging society, a surgery in geriatric patient is increasing. Patients older than 60 year are particularly affected for postoperative cognitive dysfunction (POCD) (26-41%). The patients experiencing POCD are at an increased risk of death in the first year after surgery. So, POCD is important because it can influence to patient's quality of life.

In the investigator's hospital, laparoscopic cholecystectomy is performed with increasing frequency in aging patients. So the investigator's study will be conducted in elderly patients during laparoscopic cholecystectomy. The anesthetic methods are divided into the following 3 kinds: sevoflurane, propofol, dexmedetomidine. These anesthetic drugs are used in general anesthesia generally. The control group include a spouse of the patient which must be older than 60 year and does not have anesthetic history.

After the surgery, the patients are discharged from the hospital, the investigators will check the postoperative cognitive function 4 times: 1week, 3months, 6months, 1 year later using the Korean version of telephone interview for cognitive status (TICS). The Korean version of TICS was validated tool for examination of cognitive function and this tool and mini-mental state examination (MMSE) be linked directly. The test will be administered to spouse simultaneously by telephone.

Sample size was calculated for the primary outcome parameters (whether long-term postoperative cognitive dysfunction (POCD) is occured after general anesthesia), and the investigators hypothesized that two groups are in this study, one group is for postanesthetic patients, another is for their spouses. Total sample size was calculated to 190.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years old, scheduled for laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* diseases of the central nervous system, including dementia (Mini Mental Examination Score <24),
* consumption of major tranquilizers or antidepressants
* previous neuropsychological testing
* the patient's inability to comply and follow procedures or poor comprehension of the language used in the study.
* Parkinson's disease
* Patients with a severe visual or auditory handicap, illiteracy
* alcoholism (intake of >5 units of alcohol daily during the last 3 months)
* drug dependence
* those not expected to complete the postoperative tests were excluded as well

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of long-term postoperative cognitive dysfunction after general anesthesia in elderly patients. | two years
  Investigators will assess the postoperative cognitive dysfunction after general anesthesia in elderly patients compare to spouses which have no anesthetic history. Investigators will test participants using the Korean version of TICS and test will be done 1weak, 3months, 6months, 1 year after the surgery.

SECONDARY OUTCOMES:
The difference of incidence in postoperative cognitive dysfunction after general anesthesia according to the anesthetic drugs | two years
  Investigators will assess the postoperative cognitive dysfunction (POCD) after general anesthesia (sevoflurane, propofol and dexmedetomidine) and compare the occurrence rate of the POCD in 3 anesthetic methods.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hoon Baek, Study Chair — Pusan National University Yangsan Hospital